CLINICAL TRIAL: NCT02932501
Title: International, Multicenter, Prospective Registry to Collect Data of Treatment Patterns of Patients With Medication-related Osteonecrosis of the Jaw (MRONJ) and Their Outcome
Brief Title: Medication-related Osteonecrosis of the Jaw (MRONJ) Registry
Acronym: MRONJ
Status: Active, not recruiting | Type: Observational
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Collaborators: AOCMF (Other)
Responsible Party: Sponsor
Organization: AO Innovation Translation Center (Other)
Other Study IDs: RP_MRONJ_1.0
Record Dates: First submitted 2016-10-12; First posted 2016-10-13 (Estimated); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Medication-related Osteonecrosis of the Jaw; Bisphosphonate-Associated Osteonecrosis of the Jaw
Keywords: Bisphosphonate; Jaw; Osteonecrosis; Antiresorptive drugs; Denosumab
MeSH Terms: conditions — Bisphosphonate-Associated Osteonecrosis of the Jaw; Osteonecrosis | interventions — Conservative Treatment; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MRONJ: Patients diagnosed of medication-related osteonecrosis of the jaw (MRONJ). Treatment strategies vary depending on the stage of MRONJ and can be of different nature as:
  Conservative treatment Surgical treatment Adjuvant non-surgical treatment
  Interventions: Procedure: Conservative treatment; Procedure: Surgical treatment; Procedure: Adjuvant non-surgical treatment

INTERVENTIONS:
Procedure: Conservative treatment — Disinfectant mouth rinses, Antibiotic therapy, Antifungal therapy
Procedure: Surgical treatment — Superficial debridement, Complete removal of necrotic bone, Complete bone resection, When applicable revision and soft tissue coverage
Procedure: Adjuvant non-surgical treatment — Hyperbaric oxygen therapy Pentoxifylline and tocopherol Ozone therapy Low level laser therapy Pain relief Anti-inflammatory treatment Platelet rich plasma Parathyroid hormone and teriparatide Bone morphogenetic protein

SUMMARY:
Approximately 500 patients will be included in this patient registry. Data collection includes demographics, clinical data of underlying disease and use of bisphosphonates, denosumab and antiangiogenic drugs , degree and extension of osteonecrosis, osteonecrosis-specific treatment, outcomes and complications within 1 year after treatment.

DETAILED DESCRIPTION:
Approximately 500 patients diagnosed with medication-related osteonecrosis of the jaw will be enrolled in the study. Patients will undergo standard (routine) of care treatment, either conservative or surgical or both, and followed up during one year after the initiation of the treatment. Treatment outcome (development of the condition), pain and complications will be collected and documented over the duration of the registry.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Newly diagnosed patients with osteonecrosis in a facial bone other than the jaw, or
* Newly diagnosed patients with non-exposed MRONJ (stage 0), or
* Newly diagnosed patients with exposed MRONJ, i.e:

  * Current or previous treatment with antiresorptive or antiangiogenic agents.
  * Exposed bone or bone that can be probed through an intraoral or extraoral fistula(e) in the maxillofacial region that has persisted for more than 8 weeks
  * No history of radiation therapy to the jaws or obvious metastatic diseases of the jaw
* Ability to understand the content of the patient information/ Informed Consent Form
* Willingness and ability to participate in the clinical investigation according to the Registry Plan (RP)
* Signed and dated IRB/EC-approved written informed consent
* Mental capacity to comply with post-operative regimen, evaluation and data collection

Exclusion Criteria:

* Recent history of substance abuse (i. e., recreational drugs, alcohol) that would preclude reliable assessment
* Pregnancy or women planning to conceive within the registry period
* Prisoner
* Participation in any other medical device or medicinal product study within the previous month that could influence the results of the present registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed of medication-related osteonecrosis of the jaw (MRONJ)
Sampling Method: Probability Sample
Enrollment: 518 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Treatment outcome | 6 months / 1 year
  Compared to the baseline status of the patient's condition, the outcome will be evaluated as:
  * Worsening of the osteonecrosis (e.g. size of the lesion increased)
  * No change of the osteonecrosis
  * Reduction of the osteonecrosis (e.g. size of the lesion decrease)
  * Complete mucosa healing

SECONDARY OUTCOMES:
Pain perception | 6 months / 1 year
  Numeric Rating Scale
Staging of osteonecrosis | 6 months / 1 year
  Staging of osteonecrosis according to the American Association of Oral and Maxillofacial Surgeons
Site and size of the lesion | 6 months / 1 year
  Site (single vs. multiple) and size of the lesion according to Weitzman et al.

CONTACTS AND LOCATIONS:
Overall Officials: Risto Kontio, MD DDS PhD, Principal Investigator — Helsinki University Central Hospital
Locations (14):
- University of Kentucky Chandler Medical Center, Lexington, Kentucky, United States
- Helsinki University Hospital, Helsinki, Finland
- Germany (3):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätskliniken Eppendorf, Hamburg
  - Ludwig-Maximilians University Munich, Klinik und Poliklinik für Mund-, Kiefer und Gesichtschirurgie, München
- Eramus MC, Rotterdam, Netherlands
- Hamad Medical Corporation, Doha, Qatar
- Emergency Clinical County Hospital of Constanta, Constanța, Romania
- University Medical Centre Ljubljana, Ljubljana, Slovenia
- Kyungpool National University, Daegu, South Korea
- 12 de Octubre University Hospital, Madrid, Spain
- Switzerland (3):
  - Universitätsspital Basel, Basel
  - Luzerner Kantonsspital, Lucerne
  - Universitätsspital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No